CLINICAL TRIAL: NCT02072369
Title: Simulated Home Therapy Program for the Hand After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Derek Kamper, Research Scientist, SMPP, RIC, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00032058; H133E070013, MARS (Other Grant/Funding Number: National Institute of Disability and Rehabilitation Research)
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Stroke
Keywords: stroke; hand; fingers; rehabilitation; training
MeSH Terms: conditions — Stroke | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAEDA Glove (Experimental): Voice And EMG-Driven Actuated glove used during hand occupational therapy training
  Interventions: Other: VAEDA Glove; Other: Occupational Therapy
- No-glove (Active Comparator): hand occupational therapy sessions without assistive device
  Interventions: Other: Occupational Therapy

INTERVENTIONS:
Other: VAEDA Glove — Voice And EMG-Driven Actuated glove used during training
  Arms: VAEDA Glove
Other: Occupational Therapy — novel upper extremity occupational therapy focused on the hand

SUMMARY:
The purpose of this study is to investigate the benefits of incorporating an actuated, EMG-controlled glove into occupational therapy of the hand.

DETAILED DESCRIPTION:
Stroke survivors with chronic hemiparesis of the upper extremity undertook 18 one-hour training sessions over a 6-week period. Participants received occupational therapy focusing on grasp-and-release using a task-oriented protocol developed at the Rehabilitation Institute of Chicago by Dr. Mary Ellen Stoykov. Over 90% of all repetitions performed during each session were focused on functional activities, as opposed to active exercise. The skills and strategies developed in therapy were then implemented into activities identified as goals by the participant, such as donning socks. Difficulty of the task, activity, or exercise was progressed for each participant to provide optimal challenge to enhance skill.

Subjects were assigned to one of two groups by casting lots. One group (VAEDA Glove) performed all tasks while wearing a custom Voice And EMG-Driven Actuated glove, the VAEDA Glove. The other group (No-Glove) performed the same types of tasks without use of the VAEDA Glove. The VAEDA Glove is a portable active-assistance glove, designed to assist digit extension in order to allow repeated practice of specified tasks. The glove contains cables traversing the dorsal side of the digits in order to provide extension and resist flexion. Forces are transmitted through the cables from a servomotor located remotely to the digits. The servomotor controls torque or displacement in the cable. Along the digits, the cables traverse through custom plastic blocks, which serve both to guide the cable and to prevent joint hyperextension.

The VAEDA Glove can be controlled with up to 3 channels of electromyography (EMG). For this study, electrodes were placed above flexor digitorum superficialis (FDS) and extensor digitorum communis (EDC). The group using the J-Glove could receive assistance during hand opening, but only if appropriate EMG activity was detected. The EDC EMG activity had to reach a prescribed threshold before extension assistance would be provided. Similarly, FDS EMG activity had to surpass a threshold level during hand closing before the user was allowed to flex the digits. Feedback of muscle activity was available to the user through a custom graphical user interface.

ELIGIBILITY:
Inclusion Criteria:

* chronic upper extremity hemiparesis subsequent to stroke (minimum of 6 months post-stroke)
* moderate hand impairment classified as Stage 4 on the Chedoke McMaster Stroke Assessment

Exclusion Criteria:

* anti-spasticity medications/injections taken less than 6 month prior to enrollment
* contractures greater than 20 degrees
* inability to follow single-step commands
* significant upper extremity pain (self-reported pain of greater than 6 on a 10-point scale)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The Action Research Arm Test (ARAT) | Change from Baseline after 6 weeks of training
Wolf Motor Function Test (WMFT) | Change from Baseline after 6 weeks of training
Fugl-Meyer Upper Extremity Motor Assessment (FMUE) | Change from Baseline after 6 weeks of training
Chedoke McMaster Stroke Assessment Stage of Hand (CMSA-H) | Change from Baseline after 6 weeks of training
Action Research Arm Test (ARAT) | Change from Baseline to 1 month following training completion
Wolf Motor Function Test (WMFT) | Change from Baseline to 1 month following training completion
Fugl-Meyer Upper Extremity Motor Assessment (FMUE) | Change from Baseline to 1 month following training completion
Chedoke McMaster Stroke Assessment Stage of Hand (CMSA-H) | Change from Baseline to 1 month following training completion

SECONDARY OUTCOMES:
Hand Kinematics | Change from Baseline after 6 weeks of training and 1 month follow up
  hand kinematics were measured explicitly with a CyberGlove (CyberGlove Systems LLC, San Jose, CA). From an initially relaxed, resting posture, participants were asked to extend the digits fully ("open") and then flex fully ("close") their affected hand into a fist. The CyberGlove measured joint displacement for each digit during task performance.
3-point (palmar) Pinch Strength (PPS) | Change from Baseline after 6 weeks of training and 1 month follow up
  using a pinch gauge (PG-60, B&L Engineering)
Lateral Pinch Strength (LPS) | Change from Baseline after 6 weeks of training and 1 month follow up
  using a pinch gauge (PG-60, B&L Engineering)
Grip Strength (GS) | Change from Baseline after 6 weeks of training and 1 month follow up
  JAMAR 5030J1 Hand Dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Derek G Kamper, PhD, Principal Investigator — Illinois Institute of Technology / Rehabilitation Institute of Chicago
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ochoa JM, Listenberger M, Kamper DG, Lee SW. Use of an electromyographically driven hand orthosis for training after stroke. IEEE Int Conf Rehabil Robot. 2011;2011:5975382. doi: 10.1109/ICORR.2011.5975382. PMID 22275586
- [Background] Ochoa J, Dev Narasimhan YJ, Kamper DG. Development of a portable actuated orthotic glove to facilitate gross extension of the digits for therapeutic training after stroke. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:6918-21. doi: 10.1109/IEMBS.2009.5333630. PMID 19964456